CLINICAL TRIAL: NCT05168592
Title: Exploring the Neural Mechanisms of Imaginal Extinction Using fMRI and Psychophysiology
Brief Title: The Neural Mechanisms of Imaginal Extinction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-06930b
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Fear of Spiders
Keywords: Threat conditioning; Extinction; Imaginal Extinction; Mental Imagery
MeSH Terms: conditions — Arachnophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaginal extinction (Experimental): Conditioned fear will be diminished using imaginal extinction.
  Interventions: Behavioral: Threat conditioning; Behavioral: Imaginal extinction

INTERVENTIONS:
Behavioral: Threat conditioning — Day 1: The participant is repeatedly shown two stimulus (CS+,CS-), one at a time. CS+ is paired with an electric shock. CS- acts as a control stimulus. The stimuli consist of photos of two different objects. Stimuli will be counterbalanced between participants.
Behavioral: Imaginal extinction — Day 1: Participants are repeatedly instructed to produce mental imagery of the two stimuli used during threat conditioning. Imagery is prompted through different written instructions presented in pseudo-randomized order on a screen. No shocks will be delivered.

SUMMARY:
Imaginal exposure is a widely used and effective psychological treatment technique in which patients are exposed to fearful stimuli and situations using mental imagery. This study examines imaginal extinction, an experimental analogue of imaginal exposure that allows the study of this treatment technique under controlled circumstances. During imaginal extinction, conditioned fear is diminished through repeated exposure to mental imagery of the feared (conditioned) stimulus. The neural underpinnings of imaginal extinction is not known, and hence, this study examines neural activations during imaginal extinction using psychophysiology and brain imaging.

DETAILED DESCRIPTION:
In this study, participants undergo threat conditioning to two pictures (CS+, CS-) in order to acquire a conditioned threat response. After this, the conditioned threat response is diminished through imaginal extinction (i.e extinction to the mental imagery of CS+ and CS-). Functional magnetic resonance imaging (7T) is used to measure neural activations during threat conditioning and imaginal extinction. Skin conductance is used to measure arousal response. Subjective fear and mental imagery vividness ratings will also be collected. In this way, this study aims to characterize the neural underpinnings of imaginal extinction.

Note that this study employs participants fearful of spiders. This is because data collection is shared with a related study (ClinicalTrials.gov ID 2020-06930a).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent and complete study procedures
* Fear of spiders (due to data collection together with ID 2020-06930a)

Exclusion Criteria:

* Current psychiatric disorder other than spider phobia. Current use of psychotropic medication. Current neurological conditions. MRI-contraindications (i.e metal implants in skull).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Blood oxygen level dependent contrast (BOLD-signal) during threat conditioning and imaginal extinction. | Day 1
  BOLD-signal is assessed using functional magnetic resonance imaging.
Physiological arousal response during threat conditioning and imaginal extinction. | Day 1
  Skin conductance responses are used as a measure of physiological arousal response (i.e. event-related rise in electrodermal activity to stimuli).

SECONDARY OUTCOMES:
Task-specific mental imagery vividness during imaginal extinction | Day 1
  Vividness of Imagery (scale:1-5; no image at all - image as clear and vivid as real life)
Ratings of subjective fear experienced during threat conditioning and imaginal extinction. | Day 1
  Scale 0-100; no fear at all - extreme fear
Spielberger State-Trait Anxiety Inventory (STAI-T) | One week after Day 1
  STAI-T is a self-rated questionnaire included assess trait-anxiety in the participants. Scale: 20-80, where higher scores represent higher levels of trait anxiety.
Vividness of visual imagery Questionnaire (VVIQ) | One week after Day 1
  VVIQ is used to measure individual differences in the Vividness of Visual mental Imagery; scale: 16-80 where higher scores represent a higher ability for visual imagery.

CONTACTS AND LOCATIONS:
Overall Officials: Thoma Ågren, PhD, Principal Investigator — Uppsala University
Locations (1):
- The Swedish 7T facility, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
We plan to share anonymous behavioural and brain imaging data, training material, Statistical Analysis plan, and informed consent form on the project site on Open Science Framework (https://osf.io/s54dz/).
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available from completion of analysis and publication, and onwards.
Access Criteria: Anonymous behavioural and brain imaging data, training material, and Statistical Analysis plan will be made public on the project site on Open Science Framework (https://osf.io/s54dz/)